CLINICAL TRIAL: NCT04790773
Title: Alexa, What is Eliquis and Xarelto?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to continue due to low enrollment and lack of resources.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kaman Chung, Pharmacy Manager, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001194
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Patient Engagement; Patient Satisfaction
Keywords: Technology; Patient Education
MeSH Terms: conditions — Patient Participation; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patient's will receive standard education on Xarelto and Eliquis per usual process without use of Alexa based voice recording.
- Alexa Education (Active Comparator): Patient's will opt in to receive initial education via Alexa based voice recording on Xarelto and Eliquis.
  Interventions: Other: Amazon Alexa based voice recording patient education

INTERVENTIONS:
Other: Amazon Alexa based voice recording patient education — Amazon Alexa based voice recording of medication education material
  Arms: Alexa Education

SUMMARY:
The purpose of this study is to evaluate the effectiveness of providing patient medication education about Eliquis and Xarelto through an Amazon Alexa based voice recording.

DETAILED DESCRIPTION:
Anticoagulants are considered high-risk medications due to the risk of major bleeding. The Federal Drug and Food Administration (FDA) MedWatch reporting system found that anticoagulants had the most adverse drug event (ADE) reports in 2011. Anticoagulants have also been reported as one of the leading drug classes contributing to emergency department visits3. Given the potential for serious adverse events, providing effective education to increase patient knowledge and awareness of those risks are essential. Incorporating technology into health care is becoming increasingly popular and has been shown to be effective for patient education. One reason is that technology can consistently provide complete patient education and is not subject to educator variability in providing this education.

ELIGIBILITY:
Inclusion Criteria (Patients):

* 18 years of age or older
* Have been prescribed either apixaban or rivaroxaban during their inpatient stay
* Consent to participating in the study

Inclusion Criteria (Nurses):

* Providing direct patient care in select general medicine and orthopedic surgical units
* Consent to participating in the study

Exclusion Criteria:

* Patients will be excluded if they have documented altered mental status, do not speak English, or are being prescribed rivaroxaban or apixaban on discharge only.
* Nurses will be excluded if not providing direct patient care in select general medicine and orthopedic surgical units
* Nurses declining participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
% Change in pre- and post test scores | Within 72 hours of education
  Effectiveness of Alexa based education by assessing understanding of Eliquis and Xarelto pre and post Alexa education

SECONDARY OUTCOMES:
7-day post-education retention rate | 1 week post discharge
  Assess education retention rate 7-days after initial Alexa based education performed
Nursing satisfaction | 72 hours
  Nursing satisfaction assessed by likert type scale questionnaire
  1. How satisfied are you with the Alexa anticoagulation education process compared to standard of care? Responses: Very dissatisfied - Dissatisfied - Neutral - Satisfied - Very Satisfied
  2. Do you agree or disagree that Alexa helps with your day-to-day workload? Responses: Strongly Agree - Agree - Neutral - Disagree - Strongly disagree
Patient satisfaction | 72 hours
  Patient satisfaction assessed by likert type scale questionnaire
  1. How satisfied are you with the anticoagulant education provided by Alexa? Responses: Very dissatisfied - Dissatisfied - Neutral - Satisfied - Very Satisfied
  2. How strongly would you recommend using Alexa anticoagulant education to your friends, family and/or other patients? Responses: Highly recommend - Recommend - Neutral - Do not recommend

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No